CLINICAL TRIAL: NCT00847990
Title: Non-Invasive Screening for Fetal Aneuploidy: A New Maternal Plasma Marker
Brief Title: Non-Invasive Screening for Fetal Aneuploidy
Status: Completed | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Collaborators: Obstetrix (Unknown)
Responsible Party: Sponsor
Other Study IDs: SQNM-T21-301
Record Dates: First submitted 2009-02-18; First posted 2009-02-20 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-09

CONDITIONS: Down Syndrome; Edwards Syndrome
Keywords: Down syndrome; aneuploidy; chromosome abnormality; amniocentesis; chorionic villus sampling; Laboratory Developed Test (LDT)
MeSH Terms: conditions — Down Syndrome; Trisomy 18 Syndrome; Aneuploidy; Chromosome Aberrations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — plasma, PBMCs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women who are scheduled to undergo an amniocentesis or CVS procedure and will receive the fetal FISH and/or karyotype results from the procedure.
  Interventions: Other: Maternal blood screening test for fetal aneuploidy

INTERVENTIONS:
Other: Maternal blood screening test for fetal aneuploidy — One blood draw of 20 to 30 mL

SUMMARY:
The purpose of this study is to determine if a laboratory test developed by the Sequenom Center for Molecular Medicine (SCMM) that uses a new marker found in the mother's blood can better identify pregnancies that have a child with a chromosome abnormality such as Down syndrome (Trisomy 21), Edwards syndrome (Trisomy 18), or other chromosome abnormality.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to provide written informed consent
* Pregnant female with singleton gestation 18 years of age or older
* Subject agrees to provide a 20 to 30 mL venous blood sample
* Subject is one of the following: A) currently scheduled to undergo an amniocentesis and/or CVS procedure, OR B) currently in the first trimester of pregnancy and planning to undergo an amniocentesis in the second trimester
* Subject will receive results of a genetic analysis that includes evaluation of the fetus for aneuploidy

Exclusion Criteria:

* Subject lacks the capacity to provide informed consent
* Twins, triplets or other multiple gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women who are scheduled to undergo an amniocentesis or CVS procedure and will receive the fetal FISH and/or karyotype results from the procedure.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Validate the prenatal aneuploidy LDT with blood samples from pregnant women who are undergoing invasive prenatal diagnosis | During the 1st and 2nd trimester of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Richard Porreco, MD, Principal Investigator — Obstetrix Medical Group of Colorado; Thomas J Garite, MD, Study Director — Obstetrix
Locations (25):
- United States (25):
  - Desert Good Samaritan Hospital, Mesa, Arizona
  - Banner Good Samaritan Hospital, Phoenix, Arizona
  - Phoenix Perinatal Associates, Phoenix Arizona Clinic, Phoenix, Arizona
  - Obstetric Perinatal Clinic Tucson (WOMB), Tucson, Arizona
  - Fetal Diagnostic Center, Laguna Hills, California
  - Long Beach Memorial Medical Center - Magella Medical Group, Long Beach, California
  - Obstetrix Medical Group of California - Hamilton, San Jose, California
  - Obstetrix Medical Group - Colorado at Presbyterian/St. Luke's Center, Denver, Colorado
  - Obstetrix Medical Group Colorado - Antepartum Testing Unit at Rose Medical Center, Denver, Colorado
  - Obstetrix Medical Group Colorada - Perinatal Resource Center at Swedish Medical Center, Englewood, Colorado
  - Obstetrix Medical Group - Colorado at Littleton Adventist Hospital Perinatal Care Center, Littleton, Colorado
  - Obstetrix Medical Group Colorado at Skyridge Medical Center, Lonetree, Colorado
  - Maternal Fetal Specialists - Northside Atlanta Geogia, Atlanta, Georgia
  - Maternal Fetal Specialist of John's Creek, Duluth, Georgia
  - Maternal Fetal Specialists - Gwinnett, Lawrenceville, Georgia
  - Obstetrix Medical Group of Kansas City, Missouri, Saint Luke's Perinatal Center, Kansas City, Missouri
  - Center for Maternal Fetal Medicine - 7 Hills Office, Las Vegas, Nevada
  - Center for Maternal Fetal Medicine - Pinto Office, Las Vegas, Nevada
  - Center for Maternal Fetal Medicine - Post Road Office, Las Vegas, Nevada
  - Regional Obstetrical Consultants, Chattanooga Tennessee, Chattanooga, Tennessee
  - Regional Obstetrical Consultants, Knoxville Tennessee, Knoxville, Tennessee
  - Texas Prenatal Group of San Antonio, San Antonio, Texas
  - Obstetrix Medical Group of Washington, Eastside Maternal Fetal Medicine, Bellevue, Washington
  - Obstetrix Medical Group of Washington, MFM Clinic at Evergreen Medical Center, Kirkland, Washington
  - Obstetrix Medical Group of Washington, Inc, Seattle, Washington